CLINICAL TRIAL: NCT03312530
Title: A Phase Ib/II Study of Cobimetinib Administered as Single Agent and in Combination With Venetoclax, With or Without Atezolizumab, in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of Cobimetinib Administered as Single Agent and in Combination With Venetoclax, With or Without Atezolizumab, in Participants With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO39813; 2017-000830-68 (EudraCT Number)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — cobimetinib; venetoclax; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A: Cobimetinib (Experimental): Participants will receive the standard single-agent cobimetinib dose of 60 milligrams (mg) (3 tablets of 20 mg each) orally (PO) daily on Days 1-21 of each 28-day cycle until disease progression. Upon progression, participants will be allowed to receive treatment with cobimetinib and atezolizumab at the recommended Phase II dose of cobimetinib 60 mg PO on Days 1-21 plus atezolizumab intravenous (IV) infusion at a fixed dose of 840 mg on Day 1 and Day 15 of each 28-day cycle. Treatment will continue until the participant has disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- B: Cobimetinib + Venetoclax (Experimental): Participants will receive cobimetinib PO daily on Days 1-21 of each 28-day cycle plus venetoclax PO daily on Days 1-28 of each 28-day cycle, at the dose level identified in the safety run-in phase. Treatment will continue until the participant has disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- C: Cobimetinib + Venetoclax + Atezolizumab (Experimental): Participants will receive cobimetinib PO daily on Days 1-21 of each 28-day cycle plus venetoclax PO daily on Days 1-28 of each 28-day cycle, at the dose level identified in the safety run-in phase plus atezolizumab IV infusion at a fixed dose of 840 mg on Day 1 and Day 15 of each 28-day cycle. Treatment will continue until the participant has disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax; Drug: Atezolizumab
- Safety Run-In: Cobimetinib + Venetoclax (Experimental): Participants will receive cobimetinib (on Day 1-21) plus venetoclax (on Day 1-28) at escalated doses, in 28-day cycles, to identify the dose level with acceptable safety.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax
- Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab (Experimental): Participants will receive cobimetinib (on Day 1-21) plus venetoclax (on Day 1-28) at escalated doses and atezolizumab (on Day 1 and Day 15) at a fixed dose of 840 mg IV, in 28-day cycles, to identify the dose level with acceptable safety.
  Interventions: Drug: Cobimetinib; Drug: Venetoclax; Drug: Atezolizumab

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be administered as per the schedule specified in the respective arm.
  Other Names: Cotellic®
Drug: Venetoclax — Venetoclax will be administered as per the schedule specified in the respective arm.
  Other Names: GDC-0199, ABT-199
  Arms: B: Cobimetinib + Venetoclax; C: Cobimetinib + Venetoclax + Atezolizumab; Safety Run-In: Cobimetinib + Venetoclax; Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in the respective arm.
  Arms: A: Cobimetinib; C: Cobimetinib + Venetoclax + Atezolizumab; Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab

SUMMARY:
This open-label, randomized, multicenter, triple-arm Phase Ib/II study is designed to assess the efficacy, safety, tolerability, and pharmacokinetics of cobimetinib administered as a single agent (Arm A), cobimetinib plus venetoclax (Arm B), and cobimetinib plus venetoclax plus atezolizumab (Arm C) in participants with relapsed and refractory multiple myeloma. Two successive cohorts will evaluate the safety of cobimetinib plus venetoclax and that of cobimetinib plus venetoclax plus atezolizumab in the selected population during the safety run-in phase of the study. Once the dose levels have demonstrated acceptable safety during this phase, randomization will begin for all treatment arms (Arms A, B, and C).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Documented multiple myeloma
* Received 3 to 5 prior lines of therapy for multiple myeloma, including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD)
* Achieved a response (minimal response [MR] or better) to at least one prior regimen
* Documented evidence of progressive disease (as defined by the IMWG criteria) on or after their last prior therapy, or participants who were intolerant to their last prior therapy
* Toxicities resulting from previous therapy (including peripheral neuropathy) that must be resolved or stabilized to Grade 1

Exclusion Criteria:

* Anti-myeloma treatment within 14 days or 5 pharmacokinetic (PK) half-lives of the treatment, whichever is longer, before the date of randomization
* Completion of autologous stem cell transplant within 100 days prior to the date of randomization
* Prior allogeneic stem cell transplant as well as prior solid organ transplant
* Spinal cord compression not definitively treated with surgery and/or radiation
* Prior treatment with MEK inhibitors, B-cell lymphoma-2 (Bcl-2) inhibitors, or immune checkpoint inhibitor therapies including anti-cytotoxic T-lymphocyte associated protein-4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1) or anti-programmed death-ligand 1 (anti-PD-L1)
* Treatment with systemic immunostimulatory agents within 28 days or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 14 days prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study
* Prior radiation therapy within 14 days prior to study enrollment and/or persistence of radiation-related adverse effects
* History or evidence of retinal pathology on ophthalmic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal
* History of clinically significant cardiovascular dysfunction
* Any previous venous thromboembolism greater than (>) Grade 3 within 12 months of study enrollment
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins (for participants in Arm C only)
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Active or history of autoimmune disease or immune deficiency
* History of malabsorption or other condition that would interfere with absorption of study drugs
* Active tuberculosis
* Severe infection within 28 days prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to initiation of study treatment
* Positive test results for hepatitis B (hepatitis B surface antigen [HBsAg] and/or total hepatitis B core antibody [HBcAb]) or hepatitis C virus (HCV) antibody
* Known history of human immunodeficiency virus (HIV) seropositivity
* Treatment with a live, attenuated influenza vaccine (e.g., FluMist) within 28 days prior to Cycle 1 Day 1, at any time during the study, and for at least 5 months after the last dose of study drug (for participants in Arm C only)
* Received strong cytochrome P-3A (CYP3A) inhibitors, moderate CYP3A inhibitors, strong CYP3A inducers, and moderate CYP3A inducers within 7 days prior to the initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Czechia (3):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Ostrava; Klinika hematoonkologie, Ostrava
  - Univerzita Karlova v Praze a Vseobecna fakultni nemocnice v Praze - 1; Lekarska Fakulta - I, Prague
- Denmark (2):
  - Rigshospitalet; Hæmatologisk Klinik, København Ø
  - Odense Universitetshospital, Odense C
- France (4):
  - CHU - Hôtel Dieu hematolgie clinique, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU Lyon - Centre Hospitalier Lyon Sud, Pierre-Benite (Lyon)
  - IGR, Villejuif
- Germany (4):
  - UNI-Klinikum Heidelberg Medizinische Klinik Innere Medizin V, Heidelberg
  - Uni. der Johannes Gutenberg-Universitaet Mainz; III. Medizinische Klinik und Poliklinik, Mainz
  - Universitätsklinikum Tübingen Medizinische UNI-Klinik und Poliklinik Abt. Innere Medizin II, Tübingen
  - Universtitätsklinikum Ulm; Klinik für Innere Medizin III, Ulm
- Netherlands (2):
  - Amsterdam UMC Location AMC, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (2):
  - Førde sentralsjukehus, Førde
  - Oslo University Hospital HF, Rikshospitalet, Oslo
- Poland (3):
  - Medical University School; Dept. of Haematology, Lodz
  - Uniwersytet Medyczny im.Karola Marcinkowskiego w Poznaniu, Późna
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Oncology, Warsaw
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Hematologia, Badalona, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Univ 12 de Octubre, Madrid
- Skånes Universitetssjukhus, Lund, Sweden

REFERENCES:
- [Derived] Schjesvold F, Paiva B, Ribrag V, Rodriguez-Otero P, San-Miguel JF, Robak P, Hansson M, Onishi M, Hamidi H, Malhi V, Dail M, Javery A, Ku G, Raab MS. Cobimetinib Alone and Plus Venetoclax With/Without Atezolizumab in Patients With Relapsed/Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2023 Jan;23(1):e59-e70. doi: 10.1016/j.clml.2022.10.006. Epub 2022 Oct 22. PMID 36450626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 centers in 8 countries.
Pre-assignment Details: A total of 62 participants were screened, of which a total of 49 participants were enrolled.
Groups:
- Safety Run-In: Cobimetinib + Venetoclax: Participants received cobimetinib (on Day 1-21) plus venetoclax (on Day 1-28) at escalated doses, in 28-day cycles, to identify the dose level with acceptable safety.
- Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab: Participants received cobimetinib (on Day 1-21) plus venetoclax (on Day 1-28) at escalated doses and atezolizumab (on Day 1 and Day 15) at a fixed dose of 840 mg IV, in 28-day cycles, to identify the dose level with acceptable safety.
- A: Cobimetinib: Participants received the standard single-agent cobimetinib dose of 60 milligrams (mg) (3 tablets of 20 mg each) orally (PO) daily on Days 1-21 of each 28-day cycle until disease progression. Upon progression, participants were allowed to receive treatment with cobimetinib and atezolizumab at the recommended Phase II dose of cobimetinib 60 mg PO on Days 1-21 plus atezolizumab intravenous (IV) infusion at a fixed dose of 840 mg on Day 1 and Day 15 of each 28-day cycle. Treatment continued until disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurred first.
- B: Cobimetinib + Venetoclax: Participants received cobimetinib PO daily on Days 1-21 of each 28-day cycle plus venetoclax PO daily on Days 1-28 of each 28-day cycle, at the dose level identified in the safety run-in phase. Treatment continued until disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurred first.
- C: Cobimetinib + Venetoclax + Atezolizumab: Participants received cobimetinib PO daily on Days 1-21 of each 28-day cycle plus venetoclax PO daily on Days 1-28 of each 28-day cycle, at the dose level identified in the safety run-in phase plus atezolizumab IV infusion at a fixed dose of 840 mg on Day 1 and Day 15 of each 28-day cycle. Treatment continued until disease progression, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurred first.
Period: Overall Study
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Started | 6 | 6 | 6 | 16 | 15
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 16 | 15
Not completed — Death | 5 | 5 | 4 | 10 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Participant in another sponsor study. | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 1 | 0 | 2 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Participant summarized as 'ongoing' due to missing data entry for Long-term Follow Up period on eCRF | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab | Total
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (7.6) | 66.5 (6.1) | 68.0 (5.9) | 64.1 (6.0) | 61.5 (10.5) | 64.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 6 | 3 | 18
  Male | 2 | 3 | 4 | 10 | 12 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 6 | 6 | 6 | 16 | 15 | 49
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 6 | 6 | 14 | 11 | 43
  Not Stated | 0 | 0 | 0 | 1 | 2 | 3
  Unknown | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the treatment. An AE was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. New or pre-existing conditions which worsened during the study were also considered AEs.
Time Frame: Randomization up to end of study (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15
Percentage of Participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR) as Determined by the Investigator Using International Myeloma Working Group (IMWG) Response Criteria
Description: ORR was defined as a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) and was analyzed in the safety evaluable population and in the biomarker-selected sub-populations of t(11;14) and RAS mutations.
Time Frame: From randomization to the first occurrence of a response as defined above (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15
Percentage of Participants
  Safety Population | 16.7 [0.00 to 54.82] | 33.3 [0.00 to 79.39] | 0 [0.0 to 8.33] | 31.3 [5.41 to 57.09] | 26.7 [0.95 to 52.38]
  t(11;14) Population: number analyzed (Participants) | 0 | 1 | 1 | 2 | 5
  t(11;14) Population |  | 100 [50.00 to 100.00] | 0 [0.00 to 50.00] | 100 [75.00 to 100.00] | 80.0 [34.94 to 100.00]
  RAS Mutation Population: number analyzed (Participants) | 2 | 1 | 2 | 7 | 8
  RAS Mutation Population | 0 [0.00 to 25.00] | 100 [50.00 to 100.00] | 0 [0.00 to 25.00] | 14.3 [0.00 to 47.35] | 37.5 [0.00 to 77.30]

3. Secondary Outcome: Percentage of Participants With Clinical Benefit as Determined by the Investigator Using IMWG Response Criteria
Description: Clinical benefit rate (CBR) was defined as a minimal response (MR) or better (PR,VGPR, CR, sCR).
Time Frame: From randomization to the first occurrence of disease progression or relapse or death from any cause, whichever occurs first (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15
Percentage of Participants | 33.3 [0.00 to 79.39] | 33.3 [0.00 to 79.39] | 0 [0.00 to 8.33] | 43.8 [16.32 to 71.18] | 33.3 [6.14 to 60.52]

4. Secondary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using IMWG Response Criteria
Description: PFS was defined as the time from randomization (for randomized participants) or first treatment date (for non-ranomized participants) to the first occurrence of disease progression or relapse as determined by the investigator using the IMWG criteria or death from any cause during the study, whichever occurred first.
Time Frame: From enrollment or first treatment date to the first occurrence of disease progression or relapse or death from any cause, whichever occurs first (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15
Months | 1.7 [0.9 to 3.7] | 3.4 [2.1 to 4.6] | 2.8 [1.9 to 4.7] | 4.9 [1.9 to 10.3] | 3.8 [1.4 to 4.7]

5. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using IMWG Response Criteria
Description: DOR was applicable to participants who achieved at least a PR, and was measured from the first observation of PR or better to the time of disease progression.
Time Frame: Time from the first observation of partial response (PR) or better to the time of disease progression (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 1 | 2 | 5 | 4
Months | 11.5 [NA to NA] — NA = not estimable, could not be calculated due to too few events. | 4.9 [2.3 to NA] — NA = not estimable, could not be calculated due to too few events. | 15.2 [1.9 to NA] — NA = not estimable, could not be calculated due to too few events. | NA [1.9 to NA] — NA = not estimable, could not be calculated due to too few events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization until death from any cause.
Time Frame: From randomization until death from any cause (up to approximately 3 years, 7 months)
Population: The safety evaluable population included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 6 | 6 | 16 | 15
Months | 11.4 [6.3 to 13.9] | 14.3 [14.1 to NA] — NA = not estimable, could not be calculated due to too few events. | 12.9 [3.2 to NA] — NA = not estimable, could not be calculated due to too few events. | 13.5 [8.0 to 26.9] | 22.0 [15.5 to NA] — NA = not estimable, could not be calculated due to too few events.

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Cobimetinib
Description: AUC0-24hr area under the plasma concentration-time curve from time 0 to 24 hrs
Time Frame: Pre-dose (within 1 hr), 2, 4, 6 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: The PK population included participants from Arms A, B, and C who received at least one dose of study medication and for whom at least one evaluable PK sample was collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 4 | 0 | 11 | 9
hr*ng/mL | 2390 (53.4) | 3190 (55.3) |  | 2540 (78.1) | 2900 (54.6)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cobimetinib
Description: Cmax is the maximum observed plasma concentration at steady state.
Time Frame: Pre-dose (within 1 hr), 2, 4, 6 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 0 | 13 | 12
ng/mL | 157 (63.5) | 192 (61.7) |  | 148 (72.6) | 166 (61.0)

9. Secondary Outcome: Time to Reach Cmax (Tmax) of Cobimetinib
Description: Tmax is the time to reach Cmax.
Time Frame: Pre-dose (within 1 hr), 2, 4, 6 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hr
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 0 | 13 | 12
hr | 4.00 [2.10 to 4.02] | 4.00 [2.05 to 5.73] |  | 4.00 [2.00 to 6.08] | 4.00 [2.23 to 6.37]

10. Secondary Outcome: AUClast of Venetoclax
Description: AUClast=area under the plasma concentration-time curve (samples collected to 8hr postdose on C1D15)
Time Frame: Pre-dose (within 1 hr), 2, 4, 6, 8 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: The PK population included participants from Arms B and C who received at least one dose of study medication and for whom at least one evaluable PK sample was collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 13 | 11
hr*ug/mL | 4.96 (67.2) | 5.13 (57.0) | 6.52 (63.7) | 6.52 (51.3)

11. Secondary Outcome: Cmax of Venetoclax
Description: Cmax is the maximum observed plasma concentration at steady state.
Time Frame: Pre-dose (within 1 hr), 2, 4, 6, 8 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 13 | 11
ug/mL | 1.25 (81.0) | 1.16 (48.7) | 1.32 (55.3) | 1.35 (18.2)

12. Secondary Outcome: Tmax of Venetoclax
Description: Tmax is the time to reach Cmax.
Time Frame: Pre-dose (within 1 hr), 2, 4, 6, 8 hrs post-dose on Day 15 of Cycle 1 (cycle length: 28 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 13 | 11
hr | 5.73 [3.92 to 5.77] | 5.65 [3.75 to 5.78] | 6.00 [3.95 to 8.50] | 5.92 [0 to 8.17]

13. Secondary Outcome: Percentage of Participants With Anti-Drug Antibody (ADA) to Atezolizumab
Time Frame: Pre-infusion (0 hr) on Day 1 of Cycles 1, 2, 3 (cycle length: 28 days); at treatment discontinuation visit (up to approximately 3 years, 7 months)
Population: The immunogenicity analysis population for atezolizumab consisted of all participants from Arm C with any ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | C: Cobimetinib + Venetoclax + Atezolizumab
Number analyzed (Participants) | 6 | 14
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Randomization up to end of study (up to approximately 3 years, 7 months)
Description: AEs were recorded for the safety-evaluable population, which included all participants who received any amount of study drug and analyzed according to the treatment arm they received.
Arm/Group | Safety Run-In: Cobimetinib + Venetoclax | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab | A: Cobimetinib | B: Cobimetinib + Venetoclax | C: Cobimetinib + Venetoclax + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 5/6 | 5/6 | 4/6 | 11/16 | 8/15
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 3/6 | 12/16 | 11/15
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/6 | 15/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In: Cobimetinib + Venetoclax (N=6) | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab (N=6) | A: Cobimetinib (N=6) | B: Cobimetinib + Venetoclax (N=16) | C: Cobimetinib + Venetoclax + Atezolizumab (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (2) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPHILUS SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LISTERIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 2 (2)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RESPIROVIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In: Cobimetinib + Venetoclax (N=6) | Safety Run-In: Cobimetinib + Venetoclax + Atezolizumab (N=6) | A: Cobimetinib (N=6) | B: Cobimetinib + Venetoclax (N=16) | C: Cobimetinib + Venetoclax + Atezolizumab (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 1 (1) | 9 (11) | 9 (14)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (4) | 4 (10) | 0 (0) | 2 (2) | 7 (17)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 5 (5)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLEPHARITIS (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
BLEPHAROCHALASIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHALAZION (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OPTIC NERVE CUPPING (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBRETINAL FLUID (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SWELLING OF EYELID (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 5 (10) | 6 (9) | 2 (2) | 13 (17) | 13 (21)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (7) | 4 (4) | 1 (1) | 5 (7) | 10 (11)
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 6 (10) | 3 (8)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 4 (5) | 1 (1) | 0 (0) | 3 (5) | 3 (3)
FEELING COLD (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 2 (2)
PAIN (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (5)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4)
ORAL HERPES (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMYLASE INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
BLOOD CALCIUM INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 2 (6)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (7) | 3 (5)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (3)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TROPONIN T INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
VITAMIN B12 DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (4) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AUTONOMIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPERAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BALANOPOSTHITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 5 (6)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In March 2019, this study was placed on voluntary enrollment hold. In May 2019, after an informal efficacy review, the Sponsor decided not to remove the hold and discontinued further development of the combination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03312530/Prot_SAP_000.pdf